CLINICAL TRIAL: NCT02448563
Title: Reducing Obesity in Underserved Postpartum African American Women
Acronym: RENEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Caroline Apovian, Professor of Medicine and Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-28272; R21HD061311 (NIH); U54TR001012 (NIH)
Record Dates: First submitted 2015-05-12; First posted 2015-05-19 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: Pregnancy; African American; Weight Management Program; Behavioral Modifications
MeSH Terms: conditions — Obesity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Weekly, in-person, support groups providing nutrition and physical activity education
  Interventions: Behavioral: Nutrition and physical activity education
- Control (No Intervention): Standard of care - one counseling visit with a study dietitian

INTERVENTIONS:
Behavioral: Nutrition and physical activity education — Eight weekly in-person groups
  Arms: Intervention

SUMMARY:
In this proposal, the investigators will develop a culturally-tailored, 8-week clinic-based weight loss program to reduce obesity among postpartum African American (AA) adult women that can be integrated into a postpartum care model within a clinical setting.

DETAILED DESCRIPTION:
The investigators proposal adapts The Diabetes Prevention Program (DPP) 16 session core curriculum to our 8 session model and in addition uses the cultural tailoring techniques of the DPP to address the needs of our AA population in several ways: 1) The reference materials and lesson handouts include information about the types of foods and cooking methods used by an AA culture (see Other Study Documents); 2) Topics are selected for group classes that are most appropriate for our participants such as Hip Hop or Salsa dancing for physical activity.

Participants will be randomized during the early postpartum period to either usual care or intervention. Usual care participants will be offered the weight management standard of care which is one visit with a dietitian in the Nutrition and Weight Management Center. Intervention participants will be assigned a Birth Sister for the postpartum period. They will also attend 8 weekly sessions for the weight loss program. All participants will complete study assessment visits at 6 weeks postpartum and 15 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pre-Natal:

  1. BMI greater than or equal to 25
  2. Ready to change (classified as answering yes to: Are you seriously considering trying to lose weight to reach your goal in the next 6 months?)
  3. English-speaking
* Post-partum:

  1. Live birth (based on medical record review)

Exclusion Criteria:

* Pre-Natal:

  1. Signs of moderate to severe depression based on the Patient Health Questionnaire-9 (PHQ-9)
  2. Previous enrollment in the Birth Sister's program prior to the study
* Post-partum:

  1. Signs of moderate to severe post-partum depression based on the Edinburgh Postnatal Depression Scale (EPDS)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M. Apovian, MD, Principal Investigator — Professor of Medicine and Pediatrics

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered "enrolled" when they signed the informed consent form. From the time of enrollment to intervention start, 66 participants either withdrew from the study or became lost to follow-up.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 32 (Randomized after completing Visit 2) | 30 (Randomized after completing Visit 2)
Completed | 16 | 19
Not Completed | 16 | 11
Not completed — Lost to Follow-up | 16 | 10
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention Completers: Weekly, in-person, support groups providing nutrition and physical activity education
  Nutrition and physical activity education: Eight weekly in-person groups
- Intervention Non-completers: Non-completers
  Weekly, in-person, support groups providing nutrition and physical activity education
  Nutrition and physical activity education: Eight weekly in-person groups
- Control Completers: Standard of care - one counseling visit with a study dietitian
- Control Non-completers: Non-completers
  Standard of care - one counseling visit with a study dietitian
- Total: Total of all reporting groups
Arm/Group | Intervention Completers | Intervention Non-completers | Control Completers | Control Non-completers | Total
Number analyzed (Participants) | 16 | 16 | 19 | 11 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.1) | 30.3 (7.4) | 30.5 (6.6) | 32.6 (5.3) | 30.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 19 | 11 | 62
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 16 | 19 | 11 | 62
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] | 91.4 (22.8) | 100.5 (19.8) | 92.3 (17.9) | 93.2 (12.1) | 94.3 (18.9)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.2 (8.8) | 35.6 (6.4) | 34.8 (6.1) | 34.1 (3.6) | 35.0 (6.5)
Waist circumference [Mean (Standard Deviation); unit: centimeters] | 107.3 (18.3) | 108.1 (13.8) | 109.6 (14.8) | 109.5 (8.3) | 108.6 (14.6)
Breastfeeding [Number; unit: participants]
  Yes | 12 | 12 | 13 | 4 | 41
  No | 4 | 4 | 6 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Attendance at Group Sessions and Barriers to Attendance (Logs Kept by Research Staff)
Time Frame: Weekly up to 8 weeks
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 32
participants
  Attended 75% of sessions or more | 9
  Attended at least 1 session, but <75% of sessions | 12
  Attended no sessions | 11

2. Secondary Outcome: Change From Baseline Weight to 8 Weeks
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 19
kilograms | 2.4 (0.4) | 2.2 (0.3)

3. Secondary Outcome: Participant Satisfaction as Measured by Questionnaire and Exit Interview
Time Frame: 8 weeks
Measure: Number; unit: Percentage
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 19
Percentage
  Enjoyed Program | 100 | 58
  Program met diet/exercise needs | 60 | 26
  Program met other health concerns | 73 | 32
  Interventionist was responsive to questions | 100 | 74
  Interventionist was helpful/available | 53 | 26
  Program should be continued at hospital | 93 | 58

4. Secondary Outcome: Changes in Baseline Eating Behaviors to 8 Weeks as Measured by Eating Behavior Patterns Questionnaire
Description: Items were rated on a 5 point scale (1 strongly disagree, 2 disagree, 3 neutral or not applicable, 4 agree, 5 strongly agree). We summed the scores of the component items that comprised each scale (and higher scores are those where respondents are more likely to strongly agree). What is reported in the tables are the differences in raw scores computed by subtracting the summed scores at baseline from that measured at 8 weeks (difference = 8 weeks score - Baseline score).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 19
z-score
  Low fat eating | 4.7 (2.4) | 4.2 (1.8)
  Emotional eating | 1.5 (2.0) | -1.2 (1.2)
  Snacking | -0.8 (1.3) | -2.8 (0.8)
  Cultural/lifestyle behaviors | 0.6 (1.0) | -0.6 (0.8)
  Haphazard planning | -2.3 (1.7) | -4.6 (1.1)
  Meal skipping | -1.3 (0.9) | -1.6 (0.7)

5. Secondary Outcome: Changes in Baseline Body Image to 8 Weeks as Measured by the 34-item Multidimensional Body Relations Questionnaire
Description: The Multidimensional Body Relations Questionnaire (MBSRQ-AS) includes the following subscales: Appearance Evaluation, Appearance Orientation, Overweight Preoccupation, Self-Classified Weight, and the Body Areas Satisfaction Scale (BASS). We summed the scores of the component items that comprised each scale (and higher scores are those where respondents are more likely to strongly agree). What is reported in the tables are the differences in raw scores computed by subtracting the summed scores at baseline from that measured at 8 weeks (difference = 8 weeks score - Baseline score). Scale ranges from 1-5 (1=definitely disagree, 2=mostly disagree, 3=neither agree nor disagree, 4=mostly agree, 5=definitely agree) with higher scores reflecting better outcome. A positive value shows improvement in that subscale over time.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 19
units on a scale
  Appearance evaluation | 0.1 (0.2) | 0.2 (0.1)
  Appearance orientation | -0.02 (0.1) | -0.02 (0.1)
  Body areas satisfaction | 0.1 (0.1) | 0.1 (0.1)
  Overweight preoccupation | 0.3 (0.2) | 0.1 (0.1)
  Self-classified weight | -0.1 (0.1) | -0.2 (0.1)

6. Secondary Outcome: Changes in Baseline Physical Activity to 8 Weeks as Measured by the Kaiser Physical Activity Scale
Description: Activity indices were created for each domain of activity (household/caregiving, occupational, active living, sports/exercise) by summing the domain-specific categorical responses and dividing by the number of items, giving an average value that ranged from 1 to 5. We summed the scores of the component items that comprised each scale (and higher scores are those where respondents are more likely to strongly agree). What is reported in the tables are the differences in raw scores computed by subtracting the summed scores at Baseline from that measured at 8 weeks (difference = 8 weeks score - baseline score).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 19
units on a scale
  Household/Caregiving Index | -0.1 (0.1) | 0.2 (0.1)
  Active Living Index | 0.4 (0.2) | 0.1 (0.2)
  Sports and Exercise Index | -0.6 (0.4) | -0.3 (0.3)

7. Secondary Outcome: Waist Circumference at 8 Weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Intervention Completers | Intervention Non-completers | Control Completers | Control Non-completers
Number analyzed (Participants) | 16 | 16 | 19 | 11
centimeters | 107.3 (18.3) | 108.1 (13.8) | 109.6 (14.8) | 109.5 (8.3)

ADVERSE EVENTS:
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No